CLINICAL TRIAL: NCT05476822
Title: Profiling Spike Protein Antibody Response Post COVID-19 Booster
Status: Withdrawn | Type: Observational
Why Stopped: Not submitted for IRB approval. No participants were enrolled
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nolan Hudson, Research Associate/Medical Technologist, David Grant U.S. Air Force Medical Center
Other Study IDs: FDG20210028H
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Booster; Spike Protein IgG Antibody

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults who received a full course of COVID-19 vaccine and booster: Adults at Travis Air Force Base who are Active Duty, DoD beneficiaries, and civilian employees who present with a vaccination card verifying they have received a full course of mRNA spike protein COVID vaccine (Moderna, Pfizer, or Johnson & Johnson) and booster will have antibody titers performed from blood drawn at time of enrollment, at three months, six months and nine months post vaccine booster (+/- ten days).
  Interventions: Diagnostic Test: Obtain antibody titers

INTERVENTIONS:
Diagnostic Test: Obtain antibody titers — Obtain blood samples for antibody titers at the time of enrollment, at three months, six months and nine months post vaccine booster (+/- ten days).

SUMMARY:
A descriptive study that will quantify the mean IgG antibodies remaining in vaccinated healthy participants after their COVID booster.

DETAILED DESCRIPTION:
This is primarily a descriptive study that will quantify with 95% confidence intervals the mean IgG antibodies remaining in vaccinated healthy participants three to nine months after their COVID booster. At specified intervals during this period, a titer will be performed on blood drawn from participants to quantify the IgG antibodies to the SARS-CoV-2 spike protein.

This evaluation will not be performed in a lab with CLIA certification and this study will not be used to seek an EUA from the FDA. The FDA and CLIA regulate diagnostic laboratory testing but do not regulate surveillance testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults at Travis Air Force Base who are Active Duty, DoD beneficiaries, and civilian employees who present with a vaccination card verifying they have received a full course of mRNA spike protein COVID vaccine (Moderna, Pfizer, or Johnson & Johnson) and booster.

Exclusion Criteria:

* Unvaccinated, partially vaccinated, or unable to provide proof of COVID vaccination
* Unwilling or medically unable to have an initial or follow up blood sample drawn
* Positive COVID test after receiving COVID booster
* Current history of a bleeding disorder, cancer, or are immunocompromised
* Received a COVID vaccine booster seven or more months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults at Travis Air Force Base who are Active Duty, DoD beneficiaries, and civilian employees who present with a vaccination card verifying they have received a full course of mRNA spike protein COVID vaccine (Moderna, Pfizer, or Johnson & Johnson) and booster.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Level of IgG antibody for SARS-CoV-2 spike protein at baseline (0-2.5 months post booster) | Within 2.5 months post COVID booster
  Quantify the mean IgG antibodies titers with 95% confidence interval in vaccinated healthy adult participants at baseline (0-2.5 months post COVID booster).
Level of IgG antibody for SARS-CoV-2 spike protein 3 months post COVID booster | within 3 months post COVID booster
  Quantify the mean IgG antibodies titers with 95% confidence interval in vaccinated healthy adult participants 3 months post COVID booster.
Level of IgG antibody for SARS-CoV-2 spike protein 6 months post COVID booster | within 6 months post COVID booster
  Quantify the mean IgG antibodies titers with 95% confidence interval in vaccinated healthy adult participants 6 months post COVID booster.
Level of IgG antibody for SARS-CoV-2 spike protein 9 months post COVID booster | within 9 months post COVID booster
  Quantify the mean IgG antibodies titers with 95% confidence interval in vaccinated healthy adult participants 9 months post COVID booster.

CONTACTS AND LOCATIONS:
Overall Officials: Nolan R Hudson, MS, Principal Investigator — David Grant Medical Center, Travis AFB, CA

REFERENCES:
- [Background] Thakkar A, Gonzalez-Lugo JD, Goradia N, Gali R, Shapiro LC, Pradhan K, Rahman S, Kim SY, Ko B, Sica RA, Kornblum N, Bachier-Rodriguez L, McCort M, Goel S, Perez-Soler R, Packer S, Sparano J, Gartrell B, Makower D, Goldstein YD, Wolgast L, Verma A, Halmos B. Seroconversion rates following COVID-19 vaccination among patients with cancer. Cancer Cell. 2021 Aug 9;39(8):1081-1090.e2. doi: 10.1016/j.ccell.2021.06.002. Epub 2021 Jun 5. PMID 34133951
- [Background] Kyriakidis NC, Lopez-Cortes A, Gonzalez EV, Grimaldos AB, Prado EO. SARS-CoV-2 vaccines strategies: a comprehensive review of phase 3 candidates. NPJ Vaccines. 2021 Feb 22;6(1):28. doi: 10.1038/s41541-021-00292-w. PMID 33619260
- [Background] Koczula KM, Gallotta A. Lateral flow assays. Essays Biochem. 2016 Jun 30;60(1):111-20. doi: 10.1042/EBC20150012. PMID 27365041
- [Background] Schuler CF 4th, Gherasim C, O'Shea K, Manthei DM, Chen J, Giacherio D, Troost JP, Baldwin JL, Baker JR Jr. Accurate point-of-care serology tests for COVID-19. PLoS One. 2021 Mar 16;16(3):e0248729. doi: 10.1371/journal.pone.0248729. eCollection 2021. PMID 33725025
- [Background] Karim SSA, Karim QA. Omicron SARS-CoV-2 variant: a new chapter in the COVID-19 pandemic. Lancet. 2021 Dec 11;398(10317):2126-2128. doi: 10.1016/S0140-6736(21)02758-6. Epub 2021 Dec 3. No abstract available. PMID 34871545
- [Background] Kannan SR, Spratt AN, Sharma K, Chand HS, Byrareddy SN, Singh K. Omicron SARS-CoV-2 variant: Unique features and their impact on pre-existing antibodies. J Autoimmun. 2022 Jan;126:102779. doi: 10.1016/j.jaut.2021.102779. Epub 2021 Dec 13. PMID 34915422
- [Background] Walayat S, Ahmed Z, Martin D, Puli S, Cashman M, Dhillon S. Recent advances in vaccination of non-responders to standard dose hepatitis B virus vaccine. World J Hepatol. 2015 Oct 28;7(24):2503-9. doi: 10.4254/wjh.v7.i24.2503. PMID 26523203
- [Background] CDC COVID-19 Response Team. SARS-CoV-2 B.1.1.529 (Omicron) Variant - United States, December 1-8, 2021. MMWR Morb Mortal Wkly Rep. 2021 Dec 17;70(50):1731-1734. doi: 10.15585/mmwr.mm7050e1. PMID 34914670
- See also: World-wide tracking of coronavirus cases, deaths and vaccine doses administered — https://coronavirus.jhu.edu/map.html
- See also: COVID-19 Vaccine Breakthrough Infections Reported to CDC - United States, January 1-April 30, 2021 — https://www.cdc.gov/mmwr/volumes/70/wr/mm7021e3.htm
- See also: Reduced Neutralization of SARS-CoV-2 Omicron Variant by Vaccine Sera and Monoclonal Antibodies — https://www.medrxiv.org/content/10.1101/2021.12.07.21267432v4.full-text
- See also: SARS-CoV-2 Omicron has extensive but incomplete escape of Pfizer BNT162b2 elicited neutralization and requires ACE2 for infection — https://www.ahri.org/wp-content/uploads/2021/12/MEDRXIV-2021-267417v1-Sigal.pdf
- See also: What Do We Know About the New COVID variant Omicron — https://www.cambridgeindependent.co.uk/news/what-do-we-know-about-the-new-covid-variant-omicron-9230090/
- See also: Department of Health, Government of South Africa — https://sacoronavirus.co.za/